CLINICAL TRIAL: NCT01088165
Title: The Influence of Adalimumab vs. Fumaric Acid Esters on Cardiovascular and Metabolic Risk Factors in the Therapy of Patients With Moderate to Severe Psoriasis Vulgaris
Brief Title: The Influence of Adalimumab on Cardiovascular and Metabolic Risk in Psoriasis
Acronym: CASTIP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gregor Holzer, Dr, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CASTIP1
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Psoriasis; Cardiovascular Diseases; Diabetes Mellitus, Type 2
Keywords: Psoriasis; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Adalimumab; Fumaric acid esters
MeSH Terms: conditions — Psoriasis; Cardiovascular Diseases; Diabetes Mellitus, Type 2 | interventions — Adalimumab; Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab treatment group (Experimental)
  Interventions: Drug: Adalimumab treatment arm; Other: Narrow band UVB radiation
- Fumaric acid esters treatment group (Active Comparator)
  Interventions: Drug: Fumaric acid esters treatment group; Other: Narrow band UVB radiation

INTERVENTIONS:
Drug: Adalimumab treatment arm — Adalimumab: day 1: 2x40 mg s.c., day 8: 40 mg s.c., thereafter 40 mg s.c. in biweekly intervals
  Other Names: Humira, Adalimumab
  Arms: Adalimumab treatment group
Drug: Fumaric acid esters treatment group — First week:FAE mite (DIMETHYL FUMARATE 30mg, ETHYL FUMARATE CALCIUM 87mg, ETHYL FUMARATE ZINC 3mg, ETHYL FUMARATE MAGNESIUM 5mg):day 1 and 2: 0-0-1, day 3 and 4: 1-0-1, day 5-7: 1-1-1).
  Week 2: FAE forte (DIMETHYL FUMARATE 120mg ETHYL, FUMARATE CALCIUM 87mg, ETHYL FUMARATE ZINC 3mg, ETHYL FUMARATE MAGNESIUM 5mg)starting with 0-0-1 capsule daily, thereafter weekly increases by on capsule until maximum daily dose 2-2-2. In the event of side effects (in particular, gastrointestinal disturbances or flushing) adaption of the dose (reduction or no increase) depending on the type and severity of the side effect will be performed. If remission occurs at a lower than the maximum dose that dose will be maintained throughout the rest of the study period.
  Other Names: Fumaderm
  Arms: Fumaric acid esters treatment group
Other: Narrow band UVB radiation — No reduction of 50% minimum of baseline psoriasis severity index by week 12: additional narrow band UVB radiation, 3x/week until the patients achieve PASI reduction of 75% or greater or over a maximum period of another 12 weeks.
  Initial dosage: Fitzpatrick skin phototype I and II: 0,4 J/cm2, III and IV: 0,6), 10% Increments after each radiation

SUMMARY:
Psoriasis vulgaris is no longer considered as a chronic inflammatory disease restricted to the skin. Evidence has accumulated in the past that psoriasis is a chronic inflammatory systemic disease. As in rheumatoid arthritis, the chronic inflammatory process plays a central role in the pathogenesis of associated comorbidities such as diabetes and cardiovascular disease. Since several years the armamentarium of psoriasis treatment has been broadened by the availability of TNF alpha blockers. These neutralize systemic TNF alpha which not only plays a central role in the pathogenesis of psoriasis but has also been linked to inflammatory pathways in diabetes and cardiovascular disease. While a few studies have investigated the positive effects of TNF alpha blockers on associated cardiovascular disease in rheumatoid arthritis patients, no research data exist on the effects of these therapeutic agents in patients with moderate to severe chronic plaque psoriasis.

The present study aims at determining the effects of adalimumab, a potent and frequently prescribed TNF alpha blocker for the treatment of psoriasis, on different diabetic and cardiovascular risk factors in patients receiving this treatment as a remedy for moderate to severe plaque type psoriasis. The study is designed to explore whether adalimumab is capable to prevent or modulate psoriasis-associated comorbidities by blocking systemic inflammation. The effects of adalimumab will be compared with those of fumaric acids, which represent an established traditional systemic treatment option for moderate to severe psoriasis.

Study hypothesis:

Therapy with adalimumab will lead to an improvement of several parameters that reflect the risk for diabetes and cardiovascular disease in patients with chronic plaque psoriasis due to chronic inflammation. Endothelial dysfunction, as assessed by ultrasound flow mediated dilatation, will serve as primary outcome measure. Other risk factors such as blood lipids, hsCRP, IL-6, endothelial adhesion molecules, parameters of glucose metabolism and carotid intima-media thickness will be secondary outcomes.

Aim:

If adalimumab and/or fumaric acids will show a significant impact on the above mentioned parameters, these findings would offer a new perspective for the long term management of psoriatic patients and their comorbidities.

Study design: Randomized, prospective, controlled, parallel group study

Study population: 66 patients

ELIGIBILITY:
Inclusion Criteria:

* Chronic severe plaque type psoriasis (PASI <10) requiring systemic treatment. Non-response or contraindication to previous systemic and/or light treatment
* PASI ≥ 10, BSA ≥ 10
* Age 18 - 80 years

Exclusion Criteria:

* Women of childbearing potential not taking contraceptive measures
* Pregnant or breastfeeding women
* Patients with a history or ongoing malignancy, chronic infections or autoimmune disease
* Patients with severe impairment of their general health
* Patients who are unable to understand or comply with the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
The influence of adalimumab treatment in comparison to treatment with fumaric acid esters on the functional integrity of the endothelium will be monitored by flow mediated dilatation (FMD) | 3 and 6 months

SECONDARY OUTCOMES:
The measurement of carotid artery intima-media thickness (IMT) by ultrasound will serve as a morphological substrate for evaluating the potential effect of adalimumab on signs of atherosclerosis within the vessel wall | 3 and 6 months
Influence of adalimumab in comparison to fumaric acid esters on biochemical cardiovascular and metabolic risk factors | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Tanew, MD, Principal Investigator — Medical University of Vienna Department of Dermatology
Locations (1):
- Medical University Vienna Dpt. of Dermatology, Vienna, Austria